CLINICAL TRIAL: NCT00899379
Title: A Randomized, Triple-Blind, Placebo-Controlled, Outpatient Study to Examine the Safety and Efficacy of MK462 10 mg p.o. in the Treatment of Multiple Attacks of Migraine Headache
Brief Title: Treatment of Multiple Attacks of Acute Migraine (0462-025)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-025; MK0462-025; 2009_590
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2010-07-15 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Treatment Sequence 1 (Experimental): Placebo-Rizatriptan-Rizatriptan-Rizatriptan
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: Placebo
- Treatment Sequence 2 (Experimental): Rizatriptan-Placebo-Rizatriptan-Rizatriptan
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: Placebo
- Treatment Sequence 3 (Experimental): Rizatriptan-Rizatriptan-Placebo-Rizatriptan
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: Placebo
- Treatment Sequence 4 (Experimental): Rizatriptan-Rizatriptan-Rizatriptan-Placebo
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: Placebo
- Treatment Sequence 5 (Experimental): Rizatriptan-Rizatriptan-Rizatriptan-Rizatriptan
  Interventions: Drug: rizatriptan benzoate

INTERVENTIONS:
Drug: rizatriptan benzoate — Rizatriptan 10 mg p.o. at onset of moderate to severe migraine headache
  Other Names: MK0462
Drug: Comparator: Placebo — Placebo to Rizatriptan, Oral Tablet
  Arms: Treatment Sequence 1; Treatment Sequence 2; Treatment Sequence 3; Treatment Sequence 4

SUMMARY:
A study to evaluate rizatriptan for the treatment of multiple attacks of acute migraine compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient had at least a 6-month history of migraine, with or without aura
* Patient was male, or if female must have been postmenopausal, surgically sterilized, or taking adequate contraceptive precautions.
* Patient was judged to be in good health, apart from migraine

Exclusion Criteria:

* Patient was pregnant or a nursing mother.
* Patient had abused drugs or alcohol within 12 months prior to entering the study
* Patient had a history of cardiovascular disease
* Patient had clinically significant ECG abnormality
* Patient had a resting systolic blood pressure of greater than 145 mm Hg or diastolic of less than 95 mm Hg at screening
* Patient received treatment with an investigational device or compound within 30 days of the study start
* Patient typically suffered from less then 1 or more than 8 attacks of migraine per month
* Patient had difficulty in distinguishing his/her migraine attacks from tension or interval headaches
* Patient had prior exposure to rizatriptan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 1995-04; Primary Completion 1996-01 (Actual); Study Completion 1996-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Ho TW, Rodgers A, Bigal ME. Impact of recent prior opioid use on rizatriptan efficacy. A post hoc pooled analysis. Headache. 2009 Mar;49(3):395-403. doi: 10.1111/j.1526-4610.2009.01346.x. Epub 2008 Feb 12. PMID 19222588
- [Background] Ho TW, Fan X, Rodgers A, Lines CR, Winner P, Shapiro RE. Age effects on placebo response rates in clinical trials of acute agents for migraine: pooled analysis of rizatriptan trials in adults. Cephalalgia. 2009 Jul;29(7):711-8. doi: 10.1111/j.1468-2982.2008.01788.x. Epub 2009 Feb 3. PMID 19210513
- [Result] Kramer MS, Matzura-Wolfe D, Polis A, Getson A, Amaraneni PG, Solbach MP, McHugh W, Feighner J, Silberstein S, Reines SA. A placebo-controlled crossover study of rizatriptan in the treatment of multiple migraine attacks. Rizatriptan Multiple Attack Study Group. Neurology. 1998 Sep;51(3):773-81. doi: 10.1212/wnl.51.3.773. PMID 9748025
- [Result] Block GA, Goldstein J, Polis A, Reines SA, Smith ME. Efficacy and safety of rizatriptan versus standard care during long-term treatment for migraine. Rizatriptan Multicenter Study Groups. Headache. 1998 Nov-Dec;38(10):764-71. doi: 10.1046/j.1526-4610.1998.3810764.x. PMID 11284464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 23 sites in the United States.
  First Patient Treated: April, 1995
  Last Patient Treated: January 1996
Pre-assignment Details: Patients screened at a pretreatment visit were given allocated drug supply with instructions. If by 2 months after screening, a patient still had not treated a migraine attack with test medication, he/she was to be discontinued from the study.
Groups:
- Placebo/Rizatriptan/Rizatriptan/Rizatriptan: Placebo/Rizatriptan 10 mg/Rizatriptan 10 mg/Rizatriptan 10 mg = sequence for single dose of study drug taken orally for each recurrence or new migraine (up to 4 headaches)
- Rizatriptan/Placebo/Rizatriptan/Rizatriptan: Rizatriptan 10 mg/Placebo/Rizatriptan 10 mg/Rizatriptan 10 mg = sequence for single dose of study drug taken orally for each recurrence or new migraine (up to 4 headaches)
- Rizatriptan/Rizatriptan/Placebo/Rizatriptan: Rizatriptan 10 mg/Rizatriptan 10 mg/Placebo/Rizatriptan 10 mg = sequence for single dose of study drug taken orally for each recurrence or new migraine (up to 4 headaches)
- Rizatriptan/Rizatriptan/Rizatriptan/Placebo: Rizatriptan 10 mg/Rizatriptan 10 mg/Rizatriptan 10 mg /Placebo = sequence for single dose of study drug taken orally for each recurrence or new migraine (up to 4 headaches)
- Rizatriptan/Rizatriptan/Rizatriptan/Rizatriptan: Rizatriptan 10 mg/Rizatriptan 10 mg/Rizatriptan 10 mg /Rizatriptan 10 mg = sequence for single dose of study drug taken orally for each recurrence or new migraine (up to 4 headaches)
Period: Overall Study
Arm/Group | Placebo/Rizatriptan/Rizatriptan/Rizatriptan | Rizatriptan/Placebo/Rizatriptan/Rizatriptan | Rizatriptan/Rizatriptan/Placebo/Rizatriptan | Rizatriptan/Rizatriptan/Rizatriptan/Placebo | Rizatriptan/Rizatriptan/Rizatriptan/Rizatriptan
Started | 95 (Patients who were allocated study drug) | 95 (Patients who were allocated study drug) | 95 (Patients who were allocated study drug) | 94 (Patients who were allocated study drug) | 94 (Patients who were allocated study drug)
Patients Treated | 83 (Patients who took study drug) | 82 (Patients who took study drug) | 84 (Patients who took study drug) | 77 (Patients who took study drug) | 81 (Patients who took study drug)
Patients Not Treated | 12 (Patients who did not take study drug) | 13 (Patients who did not take study drug) | 11 (Patients who did not take study drug) | 17 (Patients who did not take study drug) | 13 (Patients who did not take study drug)
Completed | 61 (Patients who took study drug and completed the study) | 66 (Patients who took study drug and completed the study) | 66 (Patients who took study drug and completed the study) | 57 (Patients who took study drug and completed the study) | 63 (Patients who took study drug and completed the study)
Not Completed | 34 | 29 | 29 | 37 | 31
Not completed — Adverse Event | 2 | 2 | 1 | 1 | 2
Not completed — Lack of Efficacy | 0 | 4 | 3 | 0 | 1
Not completed — Lost to Follow-up | 9 | 3 | 0 | 6 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 2 | 3 | 6
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 1
Not completed — Patient Uncooperative | 0 | 1 | 0 | 1 | 2
Not completed — Abnormal Baseline ECG | 0 | 0 | 0 | 1 | 0
Not completed — No Longer Met Inc/Exc Criteria | 1 | 1 | 1 | 0 | 0
Not completed — Not Completed/Entered Extn | 5 | 1 | 6 | 4 | 3
Not completed — Study Terminated | 3 | 0 | 3 | 3 | 1
Not completed — Lost to Follow-up | 3 | 1 | 0 | 2 | 5
Not completed — Withdrawal by Subject | 4 | 7 | 4 | 7 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Patient Uncooperative | 0 | 0 | 0 | 1 | 0
Not completed — Abnormal Prestudy Labs | 0 | 0 | 0 | 0 | 2
Not completed — Abnormal Baseline ECG | 0 | 0 | 1 | 1 | 0
Not completed — No Attack Pretreatment | 3 | 5 | 5 | 6 | 4
Not completed — No Longer Met Inc/Exc Criteria | 1 | 0 | 0 | 0 | 0
Not completed — Inc/Exc Criteria Not Met | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Rizatriptan/Rizatriptan/Rizatriptan | Rizatriptan/Placebo/Rizatriptan/Rizatriptan | Rizatriptan/Rizatriptan/Placebo/Rizatriptan | Rizatriptan/Rizatriptan/Rizatriptan/Placebo | Rizatriptan/Rizatriptan/Rizatriptan/Rizatriptan | Total
Number analyzed (Participants) | 83 | 82 | 84 | 77 | 81 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (9.6) | 41.0 (9.8) | 42.3 (10.6) | 39.5 (10.1) | 38.9 (10.8) | 40.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 71 | 72 | 63 | 67 | 341
  Male | 15 | 11 | 12 | 14 | 14 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 76 | 75 | 80 | 72 | 79 | 382
  Oriental | 0 | 0 | 0 | 1 | 1 | 2
  Black | 3 | 2 | 2 | 2 | 1 | 10
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Thai | 0 | 1 | 0 | 0 | 0 | 1
  Other | 3 | 3 | 2 | 2 | 0 | 10
Baseline Severity (First Attack) [Number; unit: Participants] — Each patient rated headache severity on a 4-grade scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  Participants
    Grades 0, 1: No pain, Mild, or Missing | 1 | 1 | 0 | 2 | 0 | 4
    Grade 2: Moderate | 58 | 66 | 69 | 46 | 64 | 303
    Grade 3: Severe | 24 | 15 | 15 | 29 | 17 | 100

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at 2 Hours During the First Migraine Attack Period
Description: Patients reporting pain relief defined as a reduction of headache severity from grades 2 or 3 (moderate or severe) at baseline to grades 0 or 1 (no headache or mild) at 2 hours after initial dosing for the first migraine attack
Time Frame: 2 hours
Population: The primary efficacy analysis used an all-patients-treated approach which included all patients who had at least one record of an efficacy measure after the initial dose. Missing values were imputed by carrying forward the preceding values in the same phase.
Measure: Number; unit: participants
Groups:
- Rizatriptan 10 mg: All Rizatriptan 10 mg patients from all Treatment Sequences
- Placebo: All Placebo patients from all Treatment Sequences
Arm/Group | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 320 | 82
participants
  Reporting pain relief | 246 | 30
  Not reporting pain relief | 74 | 52

2. Secondary Outcome: Pain Relief at 2 Hours During the Second Migraine Attack Period
Description: Patients reporting pain relief defined as a reduction of headache severity from grades 2 or 3 (moderate or severe) to grades 0 or 1 (no headache or mild) at 2 hours after dosing for the second migraine attack
Time Frame: 2 hours
Population: The secondary efficacy analysis used an all-patients-treated approach which included all patients who had at least one record of an efficacy measure after the initial dose. Missing values were imputed by carrying forward the preceding values in the same phase. Values were not carried forward from one attack period to the next.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 291 | 73
Participants
  Reporting pain relief | 228 | 27
  Not reporting pain relief | 63 | 46

3. Secondary Outcome: Pain Relief at 2 Hours During the Third Migraine Attack Period
Description: Patients reporting pain relief defined as a reduction of headache severity from grades 2 or 3 (moderate or severe) to grades 0 or 1 (no headache or mild) at 2 hours after dosing for the third migraine attack
Time Frame: 2 hours
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 259 | 75
Participants
  Reporting pain relief | 207 | 21
  Not reporting pain relief | 52 | 54

4. Secondary Outcome: Pain Relief at 2 Hours During the Fourth Migraine Attack Period
Description: Patients reporting pain relief defined as a reduction of headache severity from grades 2 or 3 (moderate or severe) to grades 0 or 1 (no headache or mild) at 2 hours after dosing for the fourth migraine attack
Time Frame: 2 hours
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 255 | 57
Participants
  Reporting pain relief | 190 | 31
  Not reporting pain relief | 65 | 26

ADVERSE EVENTS:
Time Frame: During the 24 hours treatment period, and up to and including 7 days after the last dose of study therapy.
Description: Although a patient may have had two or more adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
  The subjects reported at risk are subjects with follow-up after at least one dose of study drug.
Arm/Group | Rizatriptan 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/337 | 0/84
Other Adverse Events (participants affected / at risk) | 199/323 | 31/84
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 10 mg (N=323) | Placebo (N=84)
Asthenia/Fatigue (General disorders) | 17 | 0
Candidiasis (Infections and infestations) | 0 | 1
Chills (General disorders) | 0 | 1
Fever (General disorders) | 1 | 1
Pain, Abdominal (General disorders) | 5 | 0
Pain, Chest (General disorders) | 11 | 1
Palpitation (Cardiac disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1
Dry Mouth (Gastrointestinal disorders) | 11 | 1
Nausea (Gastrointestinal disorders) | 23 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Leukocytes Decreased (Blood and lymphatic system disorders) | 4 | 0
Alanine Amino Transferase (ALT) Increased (Investigations) | 4 | 0
Abnormal Sensation (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 29 | 4
Euphoria (Psychiatric disorders) | 5 | 0
Headache (Nervous system disorders) | 6 | 1
Hypesthesia (Nervous system disorders) | 2 | 1
Mental Acuity Decreased (Nervous system disorders) | 6 | 2
Nervousness (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 13 | 0
Somnolence (Nervous system disorders) | 28 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Infection, Respiratory, Upper (Infections and infestations) | 2 | 2
Flushing (Skin and subcutaneous tissue disorders) | 7 | 1
Accommodation Disorder (General disorders) | 0 | 1
Depth Perception Loss (Eye disorders) | 0 | 1
Hot Flashes (Reproductive system and breast disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Pooled Extension data for PN022- NCT00897949; PN025- NCT00899379 and PN029- NCT00897104 appears in NCT00897949

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.